CLINICAL TRIAL: NCT03750981
Title: Does High-Intensity Functional Training Improve Patient Movement and Quality of Life? A Study of CrossFit® in Cancer Survivors
Brief Title: C.A.P.A.B.L.E. (CrossFit® and Physical Activity: A Better Life Experience)
Acronym: CAPABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Beebe-Dimmer, PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-091
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cancer Survivors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A 12-week pilot intervention study introducing a high-intensi (Other)
  Interventions: Behavioral: 12 week pilot intervention study.

INTERVENTIONS:
Behavioral: 12 week pilot intervention study. — Participants will begin a 12-week high-intensity functional training program conducted at CrossFit® in the D, located in downtown Detroit, Northville Athletix in Northville and Five Lakes CrossFit® in Farmington Hills.

SUMMARY:
This study will introduce cancer survivors to cross-training with the expectation that the program proposed will ultimately result in superior improvements in functional performance, body composition and quality of life compared with the current American Cancer Society (ACS) guidelines for cancer survivors.

DETAILED DESCRIPTION:
A 12-week pilot intervention study introducing a high-intensity functional training program to 100 cancer survivors and evaluate the effects of this program on patient quality of life, functional capacity, and body composition. Response rates will be determined using various recruitment methods and estimate differences in response rates by patient characteristics including race, gender and age. Barriers to participation in the program in contacted patients who do not enroll as well as patients who enroll and do not complete the program will be described, as will participant satisfaction with enrolled participants who complete the program. The goal of this pilot study is to help refine the recruitment and program methods for a larger intervention study to test the superiority of a high-intensity interval functional training program compared with current American Cancer Society guidelines in improving functional capacity, body composition and patient reported quality of life.

Surveys will be completed by each participant weekly and physical assessments will be completed monthly.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at time of program recruitment
* Diagnosed with any cancer
* Cleared from their physician to participate in the program (We assume that most patients will have completed treatment, however if a patient is currently under treatment, this should be their oncologist. If the patient is not currently undergoing treatment, this could be primary care physician or oncologist).
* Available transportation to and from the facility on session days

Exclusion Criteria

* Widely metastatic cancers to the brain or bone may be excluded.
* Patients using mobility assistance devices may be excluded. Exclusionary criteria will be reviewed on a case-by-case basis and patients with these limitations may be included with approval from Dr. Beebe-Dimmer and the referring physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment rates | Baseline
  Enrollment rates will be calculated among those who respond to notices about the study and adherence to the program among those who enroll and to describe reported barriers to participation among respondents who do not ultimately enroll
Change in functional performance and variability in functional performance among adult cancer survivors enrolled in a high-intensity functional training program | Baseline to 12 weeks
  Physical measures of strength will be assessed by a certified trainer. To assess strength improvements deadlifts (lifting weights from floor to waist) will be performed in 10 lb. increments. A circuit will also be done with strength measures including sit ups and push ups.
Change in functional performance and variability in functional performance among adult cancer survivors enrolled in a high-intensity functional training program | Baseline to 12 weeks
  Physical measures of flexibility will be assessed by a certified trainer. To assess flexibility sit ups, squats and push up level (floor, knees, on an elevated bar, etc) will be recorded.
Change in functional performance and variability in functional performance among adult cancer survivors enrolled in a high-intensity functional training program | Baseline to 12 weeks
  Physical measures of cardiovascular strength will be assessed by a certified trainer. To assess cardiovascular strength maximum effort on a stationary bike will be recorded. Additionally, in the circuit, a maximum effort on a rowing machine will be recorded.
Change in self-reported health-related quality of life (HRQOL) and variability using the FACT questionnaire | Baseline to 12 weeks
  Quality of Life will be measured using the Functional Assessment of Cancer Therapy: General (FACT), developed by Dr. David Cella. The FACT-G is 27 items assessing physical, social/ family, emotional and functional well-being. The survey uses a five-point scale from 0 (not at all) to 4 (very much). Scoring the FACT-G is performed through a sum of item scores. Higher scores indicate a better health state.
Change in Body Composition | Baseline to 12 weeks
  Changes in weight in kg
Change in Body Composition | Baseline to 12 weeks
  Changes in body fat percentage
Change in Body Composition | Baseline to 12 weeks
  Changes in visceral fat percentage
Change in Body Composition | Baseline to 12 weeks
  Changes in muscle mass percentage
Change in Body Composition | Baseline to 12 weeks
  Changes in body mass index (BMI) - Weight and height will be combined to report BMI in kg/ m2
Change in Body Composition | Baseline to 12 weeks
  Changes in resting metabolism value
Change in Motivation | Baseline to 12 weeks
  Motivation to exercise will be collected via a survey
Satisfaction with the Program | 12 weeks
  Satisfaction with the program will be collected via a survey
Program Adherence | 12 weeks
  Program adherence will be calculated based on how many sessions each participant attended in the 13 week program, 36 session design.
Height | Baseline
  Height will be collected in meters to use in the calculation of Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Beebe-Dimmer, MPH, PhD., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No